CLINICAL TRIAL: NCT04068441
Title: Measurement for Viral Reservoir and Immune Function in HIV-1-infected Patients Under Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904090RINA
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2022-09

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sample with DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular treatment: no intervention
  Interventions: Other: no intervention
- Treatment interruption: no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
Current antiretroviral therapy (ART) is highly effective to suppress plasma viral load to below the detection limit and to restore the host immunity, thus to prolong the survival of HIV-1-infected patients remarkably. However, HIV-1 will rebound to pre-treatment levels within weeks of interruption or irregular medication. The reason why HIV-1 would not be eradicated by powerful ART can be explained by that the reservoir of latent HIV-1 in resting CD4 T cells will persistently exist even long-term suppression of plasma viral RNA. Several therapeutic approaches that aim to prevent or delay viral rebound after treatment interruption, producing a post-treatment remission or functional cure of HIV-1, are being investigated. This study is to measure the size of viral reservoir and HIV-1-specific T cell response in HIV-1-infected patients during ART to help understand the mechanism of HIV-1 persistence, then to help establish a potential policy for functional cure.

DETAILED DESCRIPTION:
Introduction

Current antiretroviral therapy (ART) is highly effective to suppress plasma viral load to below the detection limit and to restore the host immunity, thus to prolong the survival of HIV-1-infected patients remarkably. However, HIV-1 will rebound to pre-treatment levels within weeks of interruption or irregular medication1,2. The reason why HIV-1 would not be eradicated by powerful ART can be explained by that the reservoir of latent HIV-1 in resting CD4 T cells will persistently exist even long-term suppression of plasma viral RNA. Several therapeutic approaches that aim to prevent or delay viral rebound after treatment interruption, producing a post-treatment remission or functional cure of HIV-1, are being investigated3. This study is to measure the size of viral reservoir and HIV-1-specific T cell response in HIV-1-infected patients during ART to help understand the mechanism of HIV-1 persistence, then to help establish a potential policy for functional cure.

Methods Enrollment criteria

1. Confirmed HIV-1 infected patients under regular follow-up and receiving antiretroviral therapy
2. Men with 20-50 years old

Exclusion criteria

1. Serious co-morbidity
2. Obvious hepatic or renal dysfunction
3. Receiving immunosuppressive therapy

Duration and frequency A total of 48 weeks of follow-up, and laboratory measurement every 8 weeks

Laboratory measurement We will draw the blood specimen from subjects after they sign the informed consent. About 30 mL blood will be taken and sent for the determination of viral reservoir and HIV-1-specific T cell responses, every 8 weeks, from the baseline at enrollment to the end of 48 weeks.

HIV-1 Gag-specific T-cell responses Recombinant HIV-1 Gag p24 (5 ug/mL; Research Diagnostics, Inc.) will be used as HIV-1 antigen. PBMC (106) will be incubated with or without p24 in 24-well plats for 6 days. The frequency of T cells with BrdU incorporation will be measured by flow cytometry.

HIV Viral Reservoirs

Levels and contents of HIV viral reservoirs in the peripheral blood will be analyzed in CD4+ T cells(the major cell type harboring HIV reservoir) in 2 major components:

* Proviral DNA
* Cell-associated (CA) HIV RNAs The quantifications for both HIV pvDNA and CA RNAare based on the PCRbasedquantitative system.

Proviral DNA Assessment The blood samples will be used to isolate CD4+ T cells for cellular DNA extraction.

Standardized aliquot amount of extracted DNA is used to determine HIV pvDNA level throughPCR-based quantitative assay targeting the conserved region of HIV gene. The HIV pvDNAlevel will be presented as copies per million CD4+ T cells.The input cell number is determined by a separate PCR targeting human endogenous gene(s).

Cell-associated (CA) HIV RNA Total cellular RNA will be extracted from CD4+ T cells to generate totalcomplementary DNA (cDNA) through reverse transcription. The cDNA is then used to determine CA HIV RNA level through PCR-based quantitative assay that targets the conserved sequences of HIV at a designated laboratory by Sponsor. The CA RNA level is presented a scopies of endogenous house-keeping gene transcripts, whose copy number will be determined independently by a separate PCR targeting the RNA transcripts of the house-keeping gene.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1-infected patients
* 20-50 years old
* receiving antiretroviral therapy

Exclusion Criteria:

* Serious co-morbidity
* Obvious hepatic or renal dysfunction
* Receiving immunosuppressive therapy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-1 infected patients receiving antiretroviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-01-28 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Changes of Proviral DNA levels | The changes of baseline proviral DNA at 48 weeks
  quantitative proviral DNA measurement as the marker of HIV reservoir

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh SM, Pan SC, Huang YS, Chang SC. Reversal of Viral Latency and Induction of Gag-Specific T-Cell Responses in HIV-1-Infected Adults Through Cyclic Treatment Interruption of Rosuvastatin: A Proof-of-Concept Study. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):500-508. doi: 10.1097/QAI.0000000000002577. PMID 33620177